CLINICAL TRIAL: NCT01007071
Title: Effects of Growth Hormone on Cognition and Cerebral Metabolism in Adults
Brief Title: Effects of Growth Hormone on Cognition and Cerebral Metabolism in Adults With Growth Hormone Deficiency
Acronym: GHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Laurence Katznelson, Professor of Neurosurgery and Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU-10022009-4140; IRB eprotocol # 15129
Record Dates: First submitted 2009-10-30; First posted 2009-11-03 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism | interventions — somatotropin (1-134); Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth hormone (Experimental): Subjects randomized to growth hormone (1-134) for 16 weeks. In this arm, growth hormone is dosed sc on a daily basis and increased over first 6 weeks (Men: start at 0.2 mg sc/d, increase to 0.6 mg sc/d after 4 weeks. Women, postmenopausal: start at 0.3 mg sc/d, increase to 0.9 mg sc/d after 4 weeks. Dose adjustments based on serum insulin-like growth factor-1 (IGF-1) levels at 6 and 12 weeks, with final IGF-1 measurement for efficacy performed at 16 weeks, with goal in range of -0.5 standard deviation (SD) to +2SD. An elevated serum IGF-1 value will result in a 20% dose reduction in GH in an active and random placebo patient. Similarly, a low serum IGF-1 will result in a 20% dose increase in an active and random placebo subject.
  Interventions: Drug: Human Growth Hormone (1-134)
- Placebo (Placebo Comparator): Subjects randomized to placebo for 16 weeks. As noted above, placebo subjects will be initiated on a daily subcutaneous injection, with dose changes based on changes in active drug subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human Growth Hormone (1-134) — Subjects randomized to human growth hormone (1-134) for 16 weeks. In this arm, growth hormone is dosed sc on a daily basis and increased over first 6 weeks (Men: start at 0.2 mg sc/d, increase to 0.6 mg sc/d after 4 weeks. Women, postmenopausal: start at 0.3 mg sc/d, increase to 0.9 mg sc/d after 4 weeks. Women premenopausal or on estrogen: start at 0.6 mg sc/d, increase to 1.3 mg sc/d after 4 weeks.) Dose adjustments based on serum IGF-1 levels at 6 and 12 weeks, with final IGF-1 measurement for efficacy performed at 16 weeks, with goal in range of -0.5 SD to +2SD. An elevated serum IGF-1 value will result in a 20% dose reduction in GH in an active and random placebo patient. Similarly, a low serum IGF-1 will result in a 20% dose increase in an active and random placebo subject.
  Other Names: Nutropin (brand name)
  Arms: Growth hormone
Drug: Placebo — Subjects randomized to placebo
  Arms: Placebo

SUMMARY:
Patients with Growth hormone (GH) deficiency often report impaired quality of life and difficulty with mental functioning. It has been suggested that GH replacement in such patients leads to improvement in cognitive function. The aim of this study is to elucidate the effects of GH replacement in patients with GH deficiency on cognitive function using structural and functional neuroimaging and cognitive testing.

DETAILED DESCRIPTION:
Eligibility screening: Diagnosis of GHD will be based on standard testing, including a blunted GH response to stimulation with glucagon provocation, defined as GH <3 microgram/l. Subjects with adult-onset GH deficiency will be included if they are age 18-65 years old, naive to GH replacement therapy, in good general health, and on stable thyroid, glucocorticoid (at replacement doses) and gonadal replacement therapy for at least 6 weeks prior to study initiation. Patients with history a Major Depression will be excluded.

Baseline: Qualifying subjects will be admitted to the CTRU for the following: Weight, body mass index, waist/hip ratio, menstrual cycle history on female subjects and vital signs. Initial clinical laboratory assessments will include IGF-1, a complete blood count, liver function tests, free T4, and a serum pregnancy test for women. Subjects will undergo 3 hours of neuropsychological testing when attention, working memory, executive function and verbal memory will be assessed with the Wechsler Adult Intelligence Scale III and Wechsler Memory Scale (WMS III). Quality of life and mood will be quantified through the Quality of Life Scale, Hamilton Rating Scale for Depression and the Quality of Life Assessment of Growth Hormone Deficiency in Adults (Qol AGHDA). After a lunch break, the patients will undergo a 1 hour MRI scan. Resting images will be obtained, and thereafter simple letters, words or pictures will be projected to subjects while in the scanner. The subjects will be asked simple questions relating to these stimuli.

Randomization and treatment: Following completion of the baseline measurements, study participants will be randomized in a double blind fashion to receive either active treatment with GH or placebo for a period of 16 weeks. GH dosages will be increased incrementally over the first 6 weeks. At 16 weeks, all subjects randomized to placebo will be switched to GH in an open label fashion with dose schedules based on the above titration. Subjects initially randomized to GH will continue to receive GH with their endocrinologist without further follow up for the study.

For efficacy measures, neuropsychological testing and fMRI will be performed at baseline and at 16 weeks, and, for subjects initially randomized to placebo, repeat studies will be performed at 32 weeks.

Safety monitoring will include assessment of changes in thyroid and adrenal status, as well as changes in liver function.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 18-65 years old
* Both men and women
* Naive to GH replacement therapy
* Diagnosis of Growth Hormone deficiency, adult onset
* Good general health
* Normal thyroid, adrenal or gonadal function, or stable thyroid, glucocorticoid (at replacement doses) and gonadal replacement therapy for at least 3 months prior to study initiation. If subjects are receiving transdermal testosterone, attainment of mid-normal serum values will be considered adequate. If subjects are on intramuscular testosterone, attainment of mid-normal serum testosterone at mid-injection cycle will be considered adequate

Exclusion Criteria:

* Pregnancy (positive pregnancy test) prior to enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if Growth Hormone therapy was initiated
* Idiopathic Growth Hormone Deficiency
* DSM IV diagnosis of Major Depressive Disorder with or without psychotic features, Bipolar II Disorder with or without psychotic features in a major depressive episode
* Current use of psychotropic medications
* History of moderate to severe brain injury
* Clinically significant cardiovascular disease
* Anemia with hct<30
* Renal insufficiency with creatinine >2.0
* Recent history of excessive alcohol use
* Participation in another simultaneous medical investigation or trial
* Active neoplasm
* Prader Willi Syndrome
* History of brain radiation
* Chemotherapy, past or present use
* History of head or eye injury involving persistent metal fragments, and implanted electrical device (such as a heart pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2012-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Era Sidhaye Shah, Sub-Investigator — Stanford University; Laurence Katznelson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the neuroendocrine center at Stanford Hospital
Pre-assignment Details: All patients were naïve to study drug, per protocol and eligibility criteria. Therefore, no washouts or other required delays were part of the study.
Groups:
- Growth Hormone: Subjects were randomized to receive growth Human Growth Hormone (1-134) (Nutropin) for 16 weeks
- Placebo: Subjects were randomized to receive placebo for 16 weeks, and then were immediately crossed over to receive active study drug for 16 weeks
Period: Overall Study
Arm/Group | Growth Hormone | Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all subjects were adults with growth hormone deficiency based on standard definitions.
Groups:
- Growth Hormone: Subjects were randomized to receive growth Human Growth Hormone (1-134) (Nutropin) for 16 weeks
  All subjects were diagnosed with growth hormone deficiency using standard testing.
- Placebo: Subjects were randomized to receive placebo for 16 weeks, and then were immediately crossed over to receive active study drug for 16 weeks
  All subjects were diagnosed with growth hormone deficiency using standard testing.
- Total: Total of all reporting groups
Arm/Group | Growth Hormone | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: BOLD Signal Measured by Functional MRI Scan to Functional Connectivity Measured by fMRI
Description: Functional MRI scans were to be performed at baseline and at 16 weeks. Changes in functional connectivity before and after 16 weeks of treatment were analyzed. The analysis involved approximately 40,000 paired sample t-tests. The dependent variable here for each subject is the correlation between the BOLD timeseries in the seed region (posterior cingulate cortex) and the BOLD timeseries in a given, standard space, brain voxel. This paired-sample t-test is run, separately, for every voxel in the brain. The pre-specified Outcome Measure intended to report the number of voxels that showed significant changes with active treatment. A preliminary analysis was conducted using a paired-sample t-test at each of the 40,000+ voxels, however, none of the voxels reached the level of significance. Since no significant voxels were detected, subsequent planned analyses were not performed, and summary level data cannot be reported for this Outcome Measure.
Time Frame: Baseline and 16 weeks
Population: Preliminary analysis did not work as intended and subsequent data were not collected from any participants (please see the detailed explanation in the Measure Description).
Groups:
- Growth Hormone: Subjects randomized to growth hormone for 16 weeks
  Human Growth Hormone (1-134): Subjects to receive growth hormone
- Placebo: Subjects randomized to placebo for 16 weeks Placebo: Subjects randomized to placebo
Arm/Group | Growth Hormone | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Neuropsychological Testing of Executive Function
Description: Executive function was assessed in part B of the 2-part Trail Making Test. In Part A, 25 circles are distributed over a sheet of paper, numbered 1 - 25, and the patient draws lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1-13) and letters (A-L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient is instructed to connect the circles as quickly as possible. The amount of time the patient takes to connect the circles is recorded as their score. If patients make an error, they are corrected then continue from the last correct circle. The number of seconds for completion of part B is reported, therefore higher scores reveal greater impairment.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Growth Hormone | Placebo
Number analyzed (Participants) | 5 | 5
seconds | 69.4 (4.5) | 77.6 (25.5)

ADVERSE EVENTS:
Time Frame: Data were collected during study (16 weeks) and for subsequent 4 months.
Description: No difference in definition.
Groups:
- Human Growth Hormone (1-134): This arm received study drug for 16 weeks. There were no serious adverse events.
- Placebo: This arm received placebo for 16 weeks. There were no serious adverse evens in this group.
Arm/Group | Human Growth Hormone (1-134) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Growth Hormone (1-134) (N=6) | Placebo (N=5)
chest pain (Cardiac disorders) | 0 (0) | 1 (1) — Subject presented to a local emergency room with atypical chest pain. His evaluation was negative including ECG and blood testing. He was discharged home, and continued the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No